CLINICAL TRIAL: NCT01093768
Title: Effects of Prosocial Neuropeptides on Human Brain Function in Healthy Volunteers and Individuals With Autism Spectrum Disorders
Brief Title: Brain Imaging Study of Adults With Autism Spectrum Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Diagnostic
Other Study IDs: 100068; 10-M-0068
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-04-11

CONDITIONS: Autism Spectrum Disorders
Keywords: Oxytocin; Vasopressin; Autism; Amygdala; Social Cognition; Autism Spectrum Disorders; ASD; Healthy Volunteer; HV
MeSH Terms: conditions — Autism Spectrum Disorder; Diabetes Insipidus; Autistic Disorder | interventions — Oxytocin; Vasopressins

INTERVENTIONS:
Drug: Oxytocin
Drug: Vasopressin

SUMMARY:
This research study investigates the effects of oxytocin and vasopressin on brain activity in adults with Autism Spectrum Disorders using functional magnetic resonance imaging (fMRI).

Background:

- Oxytocin and vasopressin are two hormones produced in the brain. Both hormones can influence activity in brain regions such as the amygdala that are involved in social and emotional processing. There is evidence suggesting that oxytocin and vasopressin may be implicated in autism spectrum disorders (ASD).

Objectives:

-Here, we use functional magnetic resonance imaging (fMRI) to assess the effects of oxytocin and vasopressin on brain activity in adult healthy volunteers and adults with ASD.

Eligibility:

- Right-handed individuals between 18 and 40 years of age who either have been diagnosed with autism, Asperger s disorder, or Pervasive Developmental Disorder- Not Otherwise Specified (PDD-NOS), or are healthy volunteers.

Design:

* This study requires 3 outpatient visits to the NIH Clinical Center in addition to a screening visit. Each visit will last about 2.5 hours. Participants may not smoke cigarettes or drink alcohol or caffeinated beverages for 12 hours before each visit.
* During each visit, participants will receive a nasal spray that contains one of the following: oxytocin, vasopressin, or placebo. Participants will receive a different spray at each visit.
* After using the nasal spray, participants will have an MRI scan of the brain while performing tasks with social and emotional stimuli.
* After the MRI scan, participants will complete questionnaires about mood and reaction to the tasks, and will remain in the clinic until the effects of the study medication have worn off.
* Participants will be contacted 1 day after each MRI scan for follow-up purposes.

DETAILED DESCRIPTION:
Objective: The goal of this protocol, broadly stated, is to evaluate the effects of the neuropeptides oxytocin and vasopressin on the neural systems involved in social cognition and emotional processing in healthy volunteers and individuals with autism spectrum disorders (ASD).

Study population: The research participants will be adult healthy volunteers and adults with ASD (ages 18-40 years).

Design: This will be a double-blind cross-over functional magnetic resonance imaging (fMRI) study, requiring three visits in addition to a screening visit. At each visit, participants will receive an intranasal application of oxytocin, vasopressin, or placebo and will be scanned while performing social cognition tasks and tasks involving the processing of affective stimuli. Drug order will be randomized across participants in each group (healthy controls and individuals with ASD).

Outcome measures: The outcome measures will include both performance scores and reaction times (RTs) on the behavioral tasks and changes in blood oxygenation level-dependent (BOLD) activation in the brain, in both healthy volunteers and patients with ASD. Our main brain region of interest will be the amygdala.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy Controls:

Age between 18 years and 40 years.

Blood Pressure (BP) less than 140/90

Normal EKG.

Menstrual phase: Female participants will be tested only during the follicular phase of their menstrual cycle (defined as days 6-12 after the first day of the last menstrual period).

Patients:

A diagnosis of autism, Asperger s disorder, or PPD NOS.

IQ > 80.

Age between 18 years and 40 years.

Blood Pressure (BP) less than 140/90

Normal EKG.

Menstrual phase: Female participants will be tested only during the follicular phase of their menstrual cycle (defined as days 6-12 after the first day of the last menstrual period).

EXCLUSION CRITERIA:

Healthy Controls:

Impaired hearing.

Head trauma with loss of consciousness in the last year or any evidence of functional impairment due to and persisting after head trauma.

Having a known risk from exposure to high magnetic fields (e.g. participants with pace makers) or having metallic implants (e.g. braces) in the head region (likely to create artifact on the MRI scans).

Past or present psychiatric, neurological, or severe chronic medical illness. This includes the absence of substance abuse histories, learning disabilities and all DSM IV disorders. The investigators will evaluate medical histories. Potential subjects with medical conditions that are judged not to interfere with the study may be allowed to participate.

Use of medications or drugs that would interfere with study results. This includes contraceptive hormones, steroids, medications for psychiatric symptoms like anxiety or depression, stimulants, and medications for high blood pressure. Participants will be asked to tell the investigators of any medications or drugs that they are taking. The investigators will consider the drug interactions with oxytocin and vasopressin prior to study, and participants will not be able to participate in the study if the drug interactions could be dangerous.

Pregnancy or Nursing Status: Because of the risk to an unborn fetus or infant, women who are pregnant or nursing are excluded from this protocol. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each drug administration and will not be able to participate if the pregnancy test is positive.

Patients:

Impaired hearing.

Head trauma with loss of consciousness in the last year or any evidence of functional impairment due to and persisting after head trauma.

Having a known risk from exposure to high magnetic fields (e.g. participants with pace makers) or having metallic implants (e.g. braces) in the head region (likely to create artifact on the MRI scans).

A known neurological or neurogenetic condition, such as uncontrolled epilepsy, cerebral palsy, and chromosomal abnormalities.

Use of medications or drugs that would interfere with the study results (see above).

Pregnancy or Nursing Status: Because of the risk to an unborn fetus or infant, women who are pregnant or nursing are excluded from this protocol. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each drug administration and will not be able to participate if the pregnancy test is positive.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-02-19; Primary Completion 2013-04-11 (Actual); Study Completion 2013-04-11 (Actual)

PRIMARY OUTCOMES:
Changes in brain activations | 1.5 hours

SECONDARY OUTCOMES:
Performance scores and reaction time on behavioral tasks | 1.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Swedo, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adolphs R, Tranel D, Damasio H, Damasio A. Impaired recognition of emotion in facial expressions following bilateral damage to the human amygdala. Nature. 1994 Dec 15;372(6507):669-72. doi: 10.1038/372669a0. PMID 7990957
- [Background] Barberis C, Tribollet E. Vasopressin and oxytocin receptors in the central nervous system. Crit Rev Neurobiol. 1996;10(1):119-54. doi: 10.1615/critrevneurobiol.v10.i1.60. PMID 8853957
- [Background] Bartz JA, Hollander E. Oxytocin and experimental therapeutics in autism spectrum disorders. Prog Brain Res. 2008;170:451-62. doi: 10.1016/S0079-6123(08)00435-4. PMID 18655901